CLINICAL TRIAL: NCT01235910
Title: Clinical Pharmacology of Aliskiren in Combination With Cyclosporine in Cardiac Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped early due to difficulty finding patients who met I/E criteria.
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0746
Record Dates: First submitted 2010-11-03; First posted 2010-11-08 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Hypertension; Cardiac Transplantation
Keywords: Hypertension; Cardiac transplantation; Aliskiren; Cyclosporine
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Aliskiren 75 mg once daily x 2 weeks, then aliskiren 150 mg once daily x 2 weeks, if blood pressure allows
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 75 mg once daily x 2 weeks, then aliskiren 150 mg once daily x 2 weeks, if blood pressure allows
  Other Names: Tekturna (aliskiren); Neoral (cyclosporine)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the blood pressure medication, aliskiren, in heart transplant patients. In terms of safety, the investigators will evaluate the blood levels of aliskiren and determine if aliskiren alters the blood levels of the anti-rejection medication, cyclosporine, in these patients. In terms of efficacy, the investigators will determine how well aliskiren lowers blood pressure in heart transplant patients.

DETAILED DESCRIPTION:
Hypertension is a major complication following cardiac transplantation, with a prevalence of 93% at 5 years post-transplant. Post-cardiac transplant hypertension is due to multiple factors such as use of cyclosporine, chronic kidney disease, and denervation. Hypertension in this population is difficult to treat, and most patients require therapy with multiple antihypertensive agents in order to achieve adequate blood pressure control. Aliskiren, a direct renin inhibitor, is a novel antihypertensive agent with a unique mechanism of action and potent blood pressure-lowering effects. As such, aliskiren is an attractive treatment option for post-cardiac transplant hypertension. This study will characterize the pharmacokinetic drug-drug interaction profile, pharmacodynamics, and safety of aliskiren 75 mg daily (low-dose) and 150 mg daily, when given in combination with cyclosporine, in cardiac transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* 6 months or more since cardiac transplant
* Clinically stable from a transplant perspective
* Maintained on a stable immunosuppressant regimen containing cyclosporine + an antiproliferative agent (e.g., azathioprine, mycophenolate), +/- an oral steroid
* Hypertension, as defined by a seated average systolic blood pressure of ≥ 140 mm Hg and a seated average diastolic blood pressure of ≥ 90 mm Hg, based on 3 separate measurements, spaced 2 minutes apart.

Exclusion Criteria:

* Clinical instability from a cardiac transplant perspective
* Contraindications to aliskiren therapy
* Conditions that may increase the risk of aliskiren adverse effects
* Severe hypertension
* Concomitant medications known to increase or decrease aliskiren plasma exposure.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Aquilante, Pharm.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aliskiren
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized Cyclosporine Area Under the Plasma Concentration-time Curve (AUC)
Description: The study was stopped due to difficulty finding patients who met the strict inclusion criteria. Only one patient was started on the study drug. as a result we did not analyze any cyclosporine PK (e.g.(AUCs) for this study.
Time Frame: 7 days, 14 days, 30 days (End of Study)
Measure: Number; unit: ng*h/ml/mg
Arm/Group | Aliskiren
Number analyzed (Participants) | 1
ng*h/ml/mg | NA — Values are not available for this measure. Study was stopped due to difficulty finding patients meeting strict inclusion criteria. One patient was started on the study drug. Therefore, we did not analyze any aliskiren PK (e.g. AUC) in this study.

2. Secondary Outcome: Aliskiren Plasma Concentrations
Description: Maximum plasma concentration; area under the concentration-time curve, half-life, oral clearance
  The study was stopped due to difficulty finding patients who met the strict inclusion criteria. Only one patient was started on the study drug. as a result we did not analyze any PK (e.g.(AUCs) for this study.
Time Frame: 2 weeks
Measure: Number; unit: ng*h/ml/mg
Arm/Group | Aliskiren
Number analyzed (Participants) | 1
ng*h/ml/mg | NA — Values are not available for this measure. Study was stopped due to difficulty finding patients meeting strict inclusion criteria. One patient was started on the study drug. Therefore, we did not analyze any aliskiren PK (e.g. AUC) in this study.

3. Secondary Outcome: Blood Pressure
Description: The study was stopped due to difficulty finding patients who met the strict inclusion criteria. Only one patient was started on the study drug. as a result we did not analyze any blood pressure for this study.
Time Frame: 2 weeks
Measure: Number; unit: mmHg
Arm/Group | Aliskiren
Number analyzed (Participants) | 1
mmHg | NA — Values are not available for this measure. Study was stopped due to difficulty finding patients meeting strict inclusion criteria. One patient was started on the study drug. Therefore, we did not analyze any blood pressure in this study.

ADVERSE EVENTS:
Arm/Group | Aliskiren
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was stopped due to difficulty finding patients who met the strict inclusion/exclusion criteria. Only one patient was started on study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No